CLINICAL TRIAL: NCT00777478
Title: A Phase I Dose Escalation Study With Sunitinib (SutentR) in Combination With Capecitabine and Irinotecan (Capiri) in Previously Treated Patients With Advanced Colorectal Cancer
Brief Title: Capiri-sutent Phase-1 in Advanced Colo-rectal Cancer
Acronym: sutent-capiri
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCNONCO20083
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer
Keywords: Sunitinib; Capecitabine; Irinotecan; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capiri-sutent — A dose escalating study in a 3 + 3 design will be performed. At MTD dose 14 additional patients will be treated. First, the optimal dose of sunitinib in a continuous schedule will be determined, thereafter, further dose escalation of capecitabine and irinotecan will be investigated.

SUMMARY:
The primary objective of this Phase 1 study is to identify the recommended dose of capiri and of sunitinib for combination therapy subsequent phase II trials.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of colorectal cancer
* Patients should have failed one previous line of systemic treatment for advanced disease (and not more than one treatment line), either with fluoropyrimidine monotherapy or in combination with oxaliplatin and/or bevacizumab.
* No prior treatment with irinotecan or sunitinib
* Age ≥ 18 years
* WHO PS 0-1 (see Appendix 3, corresponding with Karnofsky ≥ 70% )
* Life expectancy ≥ 12 weeks
* Written informed consent

Exclusion Criteria:

* No measurable disease according to RECIST criteria.
* Prior anti-cancer therapy < 3 weeks before first dose. For cetuximab < 30 days or bevacizumab < 60 days prior to the first dose.
* Unresolved toxicity > CTC gr 1 from previous anti-cancer therapy (including radiotherapy) except for alopecia.
* Inadequate bone marrow function (Hb ≤ 5.6 mmol/L, absolute neutrophil count (ANC) ≤ 1.5 x 109/L, platelets ≤100 x 109/L)
* renal dysfunction (serum creatinine ≥ 1.5x ULN and glomerular filtration rate ≤ 50 ml/min)
* Prothrombin time (PT) and activated partial thromboplastin time (APTT) > 2x ULRR
* Hepatic dysfunction (serum bilirubin ≥ 1.5x ULN, serum transaminases ≥ 2.5 x ULN)
* Greater than +1 proteinuria on two consecutive dipsticks taken no less then 2 weeks apart unless urinary protein < 1,5 g in a 24 Hr period.
* Pregnant or lactating women
* History of clinical signs/symptoms of CNS metastases
* Previous intolerance of fluoropyrimidine therapy, known dihydropyrimidine dehydrogenase (DPD) deficiency. Known hypersensitivity to irinotecan or sunitinib of their excipients.
* No major surgery < 4 weeks prior to study entry.
* No radiotherapy < 4 weeks prior to study entry except for palliative radiotherapy at focal sites.
* Any evidence of concurrent severe or uncontrolled disease (i.e. uncontrolled hypertension, congestive heart failure, myocardial infarction < 6 months, chronic active infection, poorly regulated diabetes mellitus)
* Any previous significant cardiovascular event during previous fluoropyrimidine therapy (i.e.

myocardial ischemia or infarction, arterial thrombosis, pulmonary emboli)

* Mean Qtc with Bazetts correction > 470 msec in screening ECG, or a history with familial long QT syndrome
* Significant haemorrhage (>30 ml bleeding/episode in the last 3 months) or haemoptysis (>5 ml fresh blood in previous 4 weeks)
* History of impairment of gastrointestinal function or -disease that may significantly impair the absorption of oral drugs (i.e. uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, bowel obstruction, or inability to swallow tablets)
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Concomitant use medication that may significantly affect hepatic cytochrome P450 drug metabolizing activity by way of enzyme induction or inhibition < 2 weeks if the first dose and throughout the study period (see Appendix 2)
* Other concomitant anti-cancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-05 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | after every completed doselevel

SECONDARY OUTCOMES:
determine the safety and toxicity profile using the CTCAE criteria. | after every completed doselevel

CONTACTS AND LOCATIONS:
Overall Officials: C.M.L. van Herpen, MD, Phd, Principal Investigator — UMCN st Radboud
Locations (1):
- University Medical Center Nijmegen st Radboud, Nijmegen, Gelderland, Netherlands